CLINICAL TRIAL: NCT00776503
Title: A Phase I/II Study of Vorinostat in Combination With Low Dose Ara-C for Patients With Intermediate-2 or High Risk Myelodysplastic Syndromes
Brief Title: Vorinostat and Low Dose Cytarabine for High Risk Myelodysplasia
Acronym: GFMVOR2007
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM VOR 2007-01
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2011-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: Epigenetic; Myelodysplasia; Cytarabine
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental): Cytarabine 10mg/m2 day 1-14 Vorinostat 400mg/d day 1-(7 or 10 or 14)
  Interventions: Drug: VORINOSTAT
- A (Experimental): Cytarabine 10mg/m2 day 1-14 Vorinostat 400mg/d day 15-(21 or 24 or 28)
  Interventions: Drug: VORINOSTAT

INTERVENTIONS:
Drug: VORINOSTAT — vorinostat; 400mg once daily; increasing duration (7-10-14 days)
  Other Names: SAHA; ZOLINZA

SUMMARY:
The purpose of this study is to determine the maximum tolerated duration and schedule of oral VORINOSTAT in addition to low dose cytarabine in the treatment of Intermediate-2 and High risk myelodysplastic syndromes.

DETAILED DESCRIPTION:
This is a multi-center, open-label, non-randomized, Phase I/II study. Patients will be treated either with arm A or B dosing schedules which contain increasing durations of exposure to vorinostat. LD Ara-C will be administered once daily, subcutaneously(SC), at 10 mg/m² in Cycle 1 and escalated to 20 mg/m² daily in Cycle 2 and above for 14 out of 28 days. Oral vorinostat will be administered as 400 mg, once daily either sequentially(Arm A) or concurrently (Arm B) with LD Ara-C in Dose Level #1 for 7 days, Dose Level #2 for 10 days, or Dose Level #3 for 14 days out of each 28-day cycle. Patients who do not have disease progression and who continue to meet eligibility criteria may receive up to 3 additional 28-day cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to participate in the study:

  1. Patient has MDS including the following FAB sub-types: refractory anemia with blast excess (RAEB) ,transformed refractory anemia with blast excess (RAEB-t) and non proliferative Chronic MyeloMonocytic Leukemias (WBC below 13G/l).
  2. Patient has a IPSS score > 1. 5 (INT-2 and high risk categories).
  3. Patient must have been previously treated with demethylating agents (including Azacitidine and Decitabine) and :

     1. failed to respond or
     2. progress after treatment.
  4. Patient is male or female, and ≥ 18 years of age on day of signing informed consent.
  5. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (See Appendix 6.1).
  6. Patient has recovered from toxicities due to prior therapy (less than grade 2) except for cytopenia
  7. Patient must have adequate organ function as indicated by the following laboratory values: serum creatinine <2mg/dl; total bilirubin <2,5ULN; AST<2,5ULN, ALT<2,5ULN, PAL<5ULN
  8. Patient is known to not be refractory to platelet transfusions.
  9. Female patient of childbearing potential has a negative serum pregnancy test (β-hCG) within 72 hours prior to receiving the first dose of vorinostat and or Ara-C . Female patient is not actively breastfeeding at the time of study entry.
  10. Female patient is either post-menopausal, free from menses for > 2 years, surgically sterilized or willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from becoming pregnant throughout the study, starting with Visit 1.
  11. Male patient agrees to use an adequate method of contraception for the duration of the study. Men should be advised not to father a child while receiving vorinostat and for 1 month post study.
  12. Patient is available for periodic blood sampling, study related assessments, and appropriate clinical management at the treating institution for the duration of the study.
  13. Patient has the ability to understand and willingness to sign an informed consent form indicating the investigational nature of the study.
  14. Patient is able to swallow capsules.

Exclusion Criteria:

1. Patient had prior treatment with an HDAC inhibitor (e.g., depsipeptide or NSC-630176, MS 275, LAQ-824, PXD-101, LBH589, MGCD0103, CRA024781, etc). Patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study. Patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period.
2. Patient has been previously treated with low dose (20 mg/m2 SC daily) Ara-C for MDS within 3 months of beginning this study.
3. Patient has active and uncontrolled infection
4. Patient has uncontrolled intercurrent illness or circumstances that could limit compliance with the study, including but not limited to the following: symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, pancreatitis, or psychiatric or social conditions that may interfere with patient compliance.
5. Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drug.
6. Patient has known human immunodeficiency virus (HIV) infection or HIV-related malignancy.
7. Patient has clinically active hepatitis B or hepatitis C infection.
8. Patient has a known allergy or hypersensitivity to any component of vorinostat or Ara-C.
9. Patient with a "currently active" second malignancy, other than nonmelanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled. Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >5 years or are considered by their physician to be at less than 30% risk of relapse.
10. Patient has received growth factors such as epoetin alfa (EPO) or granulocyte colony-stimulating factor (G-CSF) or has received non cytotoxic agents (including low dose oral chemotherapy) in the 30 days before inclusion. In case of previous cytotoxic treatment, an interval of 3 months is required.
11. Patient is on any systemic steroids that have not been stabilized to the equivalent of ≤ 10 mg/day prednisone during the 4 weeks prior to the start of the study drugs
12. Patients with clinical evidence of CNS leukemia.
13. Patient has a history of GI surgery or other procedures that might interfere with the absorption or swallowing of the study drugs.
14. Patient is unable to take and/or tolerate oral medications on a continuous basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum tolerated dose of the association | After 1 cycle of treatment

SECONDARY OUTCOMES:
To determine the clinical activity of this association | after 3 cycles of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas PREBET, MD, Principal Investigator — Groupe Francophone des Myelodysplasies; Norbert VEY, MD, Study Director — Groupe Francophone des Myelodysplasies
Locations (14):
- France (14):
  - Hôpital de la Durance, Avignon
  - Hopital Avicenne, Bobigny
  - CH René Dubos, Cergy-Pontoise
  - Hematology Dpt, Hôpital Sud Francilien, Corbeil-Essonnes
  - CHU Grenoble, Grenoble
  - Hôpital Edouard Heriot, dpt Hématologie Clinique, Lyon
  - Hematology Dpt, Institut Paoli Calmettes, Marseille
  - Hematology Dpt, Hopital de l'Hotel Dieu, Nantes
  - Hematology Dpt, Hopital Saint Louis, Paris
  - Hematology Dpt, Hopital Cochin, Paris
  - Centre Henri Bequerel, Rouen
  - Centre René Huguenin, Saint-Cloud
  - Hematology Dpt, Hopital Haute Pierre, Strasbourg
  - Hematology Dpt, Hopital Purpan, Toulouse

REFERENCES:
- [Derived] Prebet T, Braun T, Beyne-Rauzy O, Dreyfus F, Stammatoullas A, Wattel E, Ame S, Raffoux E, Delaunay J, Charbonnier A, Ades L, Fenaux P, Vey N. Combination of vorinostat and low dose cytarabine for patients with azacitidine-refractory/relapsed high risk myelodysplastic syndromes. Leuk Res. 2014 Jan;38(1):29-33. doi: 10.1016/j.leukres.2013.07.023. Epub 2013 Aug 13. PMID 23953882